CLINICAL TRIAL: NCT02361671
Title: Ultrasonographic Assessment of the Optic Nerve Sheath Diameter in Patients With Intracranial Pathology
Brief Title: Optic Nerve Sheath Diameter in Patients With Intracranial Pathology
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-8172
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Elevated Intracranial Pressure (ICP)
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optic Nerve Sheath Diameter using an ultrasound — Optic nerve sheath diameter will be measured by ultrasound preoperatively on the day of surgery, Immediate postoperative period (within 24 hours) or 6-8 weeks after surgery on the follow-up visit.

SUMMARY:
Elevated intracranial pressure (ICP) is a common and potentially life threatening condition arising from a variety of pathological conditions. The ability to monitor ICP is a crucial aspect in the management of these patients. Currently, the diagnosis of whether ICP is elevated or not is determined either with clinical signs (headache, nausea and vomiting or visual disturbances) or from the changes in the preoperative neuroimaging modalities such as computerized tomography (CT scan) and/or magnetic resonance imaging (MRI).

Recently, transorbital ultrasonography has gained popularity as a noninvasive bedside exam that has been shown to be useful in the diagnosis of raised ICP by evaluating the change in the optic nerve sheath diameter (ONSD).

The aim of our study is to use transorbital ultrasound to evaluate ONSD changes in patients with intracranial pathology and to compare the changes in the ONSD before and after surgical intervention as well as between patients with and without clinical or radiological signs of increased ICP.

DETAILED DESCRIPTION:
Elevated intracranial pressure (ICP) is a common and potentially life threatening condition arising from a variety of pathological conditions. The ability to monitor ICP is a crucial aspect in the management of these patients. Currently, the diagnosis of whether ICP is elevated or not is determined either with clinical signs (headache, nausea and vomiting or visual disturbances) or from the changes in the preoperative neuroimaging modalities such as computerized tomography (CT scan) and/or magnetic resonance imaging (MRI).

Recently, transorbital ultrasonography has gained popularity as a noninvasive bedside exam that has been shown to be useful in the diagnosis of raised ICP by evaluating the change in the optic nerve sheath diameter (ONSD).

The aim of our study is to use transorbital ultrasound to evaluate ONSD changes in patients with intracranial pathology and to compare the changes in the ONSD before and after surgical intervention as well as between patients with and without clinical or radiological signs of increased ICP.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial pathology patients scheduled for elective or emergency surgery.
* American Anesthesiologist Society physical status classification system (ASA) 1-4

Exclusion Criteria:

* history of Glaucoma,
* previous retinal surgery,
* optic neuritis,
* lack of informed consent,
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intracranial pathology patients scheduled for elective or emergency surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter, as measured by ultrasound of the optic nerve" | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dinsmore Michael, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada